CLINICAL TRIAL: NCT04372888
Title: Examining Choice Architecture for Genetic Testing Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20.205.01e
Record Dates: First submitted 2020-04-28; First posted 2020-05-04 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Decision Making

STUDY DESIGN:
Intervention Model Description: Randomization to 1 of 6 decision frames for two disease testing scenarios (arms)
Who Masked: Participant
Masking Description: participants are blinded to arm and decision frame
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rare genetic disease (Other): Hypothetical scenario 1: rare, life-altering genetic condition (congenital hypogonadotropic hypogonadism)
  Interventions: Behavioral: choice decision frame; Behavioral: opt-in decision frame; Behavioral: opt-out decision frame; Behavioral: enhanced choice (context) decision frame; Behavioral: enhanced choice (norms) decision frame; Behavioral: enhanced choice (affect) decision frame
- common genetic disease (Other): Hypothetical scenario 2: common, life-threatening genetic condition (hereditary breast and ovarian cancer)
  Interventions: Behavioral: choice decision frame; Behavioral: opt-in decision frame; Behavioral: opt-out decision frame; Behavioral: enhanced choice (context) decision frame; Behavioral: enhanced choice (norms) decision frame; Behavioral: enhanced choice (affect) decision frame

INTERVENTIONS:
Behavioral: choice decision frame — active choice for genetic testing
Behavioral: opt-in decision frame — "gain" frame for genetic testing
Behavioral: opt-out decision frame — "loss" frame for genetic testing
Behavioral: enhanced choice (context) decision frame — consequences of genetic testing
Behavioral: enhanced choice (norms) decision frame — social norms for genetic testing
Behavioral: enhanced choice (affect) decision frame — commitments for genetic testing

SUMMARY:
The goal of this application is to gain a deeper understanding of decision-making for genetic testing and identify effective choice-architecture-based strategies to improve decisions in genetic testing. The investigators hypothesize that choice architecture (i.e. framing) affects decision-making for hypothetical genetic testing scenarios.

DETAILED DESCRIPTION:
After providing opt-in electronic consent, eligible consented participants will be randomized to one of two hypothetical genetic testing scenarios (rare, life-altering genetic condition or common, life-threatening genetic condition). The genetic testing scenarios include brief detailed information about genetic testing (i.e. how results may influence treatment decisions) as well as information about standard approaches to treatment. Subjects will be randomized to receive a framing conditions (e.g. choice, opt-in, opt-out, enhanced choice). Participants will select a preferred testing option to the hypothetical scenario and will complete several validated instruments.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (18-64 yrs) residing in North America (who are members of the Amazon Mechanical Turk platform)

Exclusion Criteria:

* age <18yrs or >65yrs or residing outside of North America

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1012 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Genetic testing decision | after reading the scenario and viewing frame (approximately 10 minutes)
  Opting "yes" for genetic testing or "no" refusing genetic testing
Satisfaction with Decision Scale (SWD) | study completion (approximately 30 minutes)
  SWD is a validated 6-item instrument, items are scored on a 1-5 scale with higher scores indicating greater satisfaction with the decision taken
Decisional Regret Scale (DRS) | study completion (approximately 30 minutes)
  DRS is a validated 5-item instrument, items are scored on a 1-5 scale with higher scores indicating more regret with the decision taken

SECONDARY OUTCOMES:
Newest Vital Sign (NVS) | study completion (approximately 30 minutes)
  NVS is a validated 6-item instrument, questions are based on reading and interpreting a food label, higher scores (more correct answers) indicate greater levels of literacy and numeracy abilities
Experience with genetic disease | Baseline (study onset)
  Single "yes"/"no" question to determine a personal or family experience the genetic condition being presented in the scenario (arm)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Dwyer, PhD, Principal Investigator — Boston College
Locations (1):
- Boston College, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dwyer AA, Shen H, Zeng Z, Gregas M, Zhao M. Framing Effects on Decision-Making for Diagnostic Genetic Testing: Results from a Randomized Trial. Genes (Basel). 2021 Jun 20;12(6):941. doi: 10.3390/genes12060941. PMID 34202935